CLINICAL TRIAL: NCT00602784
Title: Double Blind, Randomized, Multicenter, Phase II Study of Immunization With a Hepatitis C Virus (HCV) Antigen Peptide Vaccine Together With Polyarginine, HCV Peptide Vaccine Alone, or Polyarginine Alone, in Patients With Chronic HCV Having Not Responded to or Relapsed From Primary Standard HCV Therapy
Brief Title: Phase II Study of Immunization With a Hepatitis C Virus (HCV) Antigen Peptide Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC41-201
Record Dates: First submitted 2008-01-04; First posted 2008-01-28 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- IC41-B-01/02 (Experimental): peptide dose 0.00 mg, polyarginine dose 2.00 mg
  Interventions: Biological: IC41
- IC41-C-01/02 (Experimental): peptide dose: 5.00 mg, polyarginine dose: 0.00 mg
  Interventions: Biological: IC41
- IC41-G-01/02 (Experimental): peptide dose: 2.50 mg, polyarginine dose: 1.25 mg
  Interventions: Biological: IC41
- IC41-H-01/02 (Experimental): peptide dose: 2.50 mg, polyarginine dose: 2.00 mg
  Interventions: Biological: IC41
- IC41-K-01/02 (Experimental): peptide dose: 5.00 mg, polyarginine dose: 2.00 mg
  Interventions: Biological: IC41

INTERVENTIONS:
Biological: IC41

SUMMARY:
The objectives are

1. to determine the immunological profile (CD4+, CD8+ cells, DTH) induced by immunization with HCV antigen peptide vaccine with polyarginine.
2. to document virological (HCV-RNA) and biochemical (ALT) responses following immunization with HCV antigen peptide vaccine with polyarginine.
3. to assess the safety of immunization with HCV antigen peptide vaccine with polyarginine.

DETAILED DESCRIPTION:
This is a double blind, randomized, parallel group, controlled, multicenter phase II study.

60 patients will be enrolled and assigned to one of the 5 dose or control groups. Each study group will include 8 patients.

Each patient will receive a total of 6 injections according to the dose of the assigned study group. The injections will be administered subcutaneously in the upper arm once every four weeks for 5 months, i.e. at days 1, 29, 57, 85, 113 and 141.

The volume of each injection will be 0.5 ml in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hepatitis C
* Non-response to or relapse from primary standard HCV therapy
* HLA A2 positive
* HCV-RNA positive
* HCV antibodies positive
* Liver biopsy within 30 months prior to inclusion
* Hematology and biochemistry laboratory results within the limits normally expected for the patient population (liver values maximal 5 times the upper limit of normal)
* Male and female
* From 18 to 65 years
* Written informed consent obtained prior to study entry

Exclusion Criteria:

* Any degree of liver cirrhosis or fibrosis of Ishak score ≥ 4 (for grading table, see APPENDIX 2: The Ishak Modified Hepatic Activity Index (HAI))
* Any liver disease other than hepatitis C
* History of autoimmune disease
* Immunodeficiency including post-organ-transplantation
* HIV infection
* Immunosuppressive therapy
* Any acute infections within 4 weeks prior to inclusion
* History of severe hypersensitivity reactions, anaphylaxis or atopy
* Diabetes mellitus, severe cardiopulmonary disorders, history of malignancy in the past 5 years
* Active or passive vaccination within 2 months prior to enrolment, and concomitant vaccination throughout the study period
* Pregnancy or lactation
* Unreliable contraception
* Alcohol consumption
* Drug abuse or addiction within 12 months prior to inclusion
* Participation in a methadone program
* Participation in another study within 1 month prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-11; Primary Completion 2004-05 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Immunological assays | study duration

SECONDARY OUTCOMES:
Safety | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Erich Tauber, M.D., Study Director — Valneva Austria GmbH